CLINICAL TRIAL: NCT04160481
Title: A Randomised, Double-blinded, Cross-over, Placebo- Controlled Pilot Study to Investigate the Effect of Tomato Extract on TMAO in Overweight or Obese Adults
Brief Title: A Pilot Study to Investigate the Effect of Water-soluble Tomato Extract on TMAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018-08-07-RESV
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Risk Factor
Keywords: gut microbiome; carciovascular risk factor

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tomato extract (Active Comparator)
  Interventions: Dietary Supplement: FruitFlow
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: FruitFlow — 300mg tomato extract
  Arms: Tomato extract
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
To determine the effect of 4 weeks daily consumption of Fruitflow on changes in plasma levels of fasting Trimethylamine N-oxide concentrations (TMAO)

DETAILED DESCRIPTION:
Tomatoes contain a range of polyphenols that are of low bioavailability and reach the colon. Data from animal studies suggest that certain polyphenols are extensively metabolized by the gut microbiota which may impact bioactivity including TMA/TMAO production. It was previously shown that a polyphenol-rich cranberry extract attenuated diet-induced metabolic syndrome in mice in a gut microbiota-dependent manner. In another mouse study the polyphenol resveratrol attenuated TMAO-induced atherosclerosis by decreasing TMAO levels and increasing hepatic bile acid neosynthesis via gut microbiota remodelling. However, human studies on polyphenol effect on TMAO levels and the gut microbiome are sparse. In a recent study TMAO serum levels were reduced in healthy subjects upon supplementation with a grape pomace polyphenolic extract.

This clinical study will provide new insight into the effect of tomato extract on TMAO levels and the gut microbiota composition and thus potential new mechanisms responsible for the cardiovascular protective effects.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent;
2. Be between 35 and 65 years of age;
3. Has a BMI between 28 - 35 Kg/m2;
4. Has a stable body weight (≤5% change) over the past 3-months;
5. Is in general good health, as determined by the investigator;
6. Avoid consuming dietary supplements (prebiotic, probiotic, fibre, resveratrol, fish oil, seed oils, ginkgo biloba, ginseng, fruit powder extracts and DHA) within 4 weeks prior to baseline visit, until the end of the study;
7. Avoid consuming seafood or fish 24h prior to each visit;
8. Maintain current level of physical activity;
9. Willing to consume the investigational product daily for the duration of the study.

   Exclusion Criteria:
10. Pregnant or breastfeeding women; women planning to become pregnant during the study;
11. Are hypersensitive to any of the components of the test product;
12. Has taken antibiotics within the previous 3 months;
13. Has taken hypolipidemic agents or any treatment for diabetes (type I or II) within the previous 6 months;
14. Has a history of drug and/or alcohol abuse at the time of enrolment;
15. Consumes greater than 2 servings/day of alcohol (e.g. >28 g ethanol/day);
16. Is a smoker;
17. Has made any major dietary changes in the past 3 months;
18. Planned major changes in life style (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
19. Has an eating disorder;
20. Is vegetarian/vegan diet or has food allergies or other issues with foods that would preclude intake of the study products;
21. Is using fibre supplements or enemas;
22. Has any health conditions that would prevent from fulfilling the study requirements, put the subject at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results;
23. Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney or liver disease, gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease or any condition which contraindicates, in the investigator's judgement, entry to the study;
24. Current hepatic failure, renal failure, bleeding disorder (haemophilia, Von Willebrand disease, oesophageal varicoses);
25. Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include Statins (including atorvastatin (Lipitor and Torvast), fluvastatin (Lescol), lovastatin (Mevacor, Altocor, Altoprev), pitavastatin (Livalo, Pitava), pravastatin (Pravachol, Selektine, Lipostat), rosuvastatin (Crestor) and simvastatin (Zocor, Lipex)), Cholesterol Absorption Inhibitors (including Zetia (ezetimibe)), Niacin (nicotinic acid), Fibric acid derivatives (including Atromid-S (clofibrate), Lopid (gemfibrozil), and Tricor (fenofibrate)), Bile Acid Sequestrants (including cholestyramine, sold under the brand names Questran, Prevalite, and LoCholest, and colestipol (Colestid)) or have taken them in the past 28 days;
26. Taking a cholesterol lowering supplement, including, example Plant sterols/stanols, Fish Oil supplements, vitamin B supplements (e.g. Niacin and Niacinamide), red rice yeast extract, oat beta glucan, pharmaceutical garlic or have taken them in the past month;
27. Has an active gastrointestinal disorder or previous gastrointestinal surgery;
28. If taking chronic medications (e.g., anti-hypertensive medications), they must have been taking the product for at least two months prior to screening and agree to maintain the same dosage throughout the study;
29. Has a gastrointestinal or chronic infective disease (i.e., diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.), with a history of such diseases;
30. Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year);
31. Experiences alarm features such as weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
32. Have a malignant disease or any concomitant end-stage organ disease;
33. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
34. Subjects may not be receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study;
35. High habitual intake of tomatoes, and tomato-based products confirmed by FFQ.
36. Known history of allergies to tomatoes or tomato-based products;

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in TMAO concentrations | 4 weeks
  Changes in plasma levels of fasting Trimethylamine N-oxide concentrations (TMAO) at baseline.

SECONDARY OUTCOMES:
Changes in the relative abundance of common human gut microbes in stool samples | 4 weeks
  Bifidobacterium sp. Blautia sp. Clostridium sp. Collinsella sp. Dorea sp. Eubacterium sp. Faecalibacterium prausnitziiLachnospira sp. Lactobacillus sp. Parabacteroides sp. Akkermansia Roseburia sp. Ruminococcus sp. Streptococcus sp. Bacillus sp. E. coli PseudomonasStaphylococcus sp. Bacteroides fragilis Salmonella sp. Shigella sp.Campylobacter sp. Yersinia sp
Urinary TMAO | 4 weeks
  Changes in urine levels of fasting TMAO
LPS | 4 weeks
  Changes in plasma levels of lipopolysaccharide (LPS)
Stool consistency | 4 weeks
  Changes in stool consistency as determined by the Bristol Stool Scale Stool Chart (BSC)
Stool microbiota composition alpha diversity | 4 weeks
  Changes in total (DNA) and active (RNA) microbiome in stool as measured by: Observed number of taxa, Shannon index of diversity, Chao I, ACE, Evenness
Stool microbiota composition beta diversity | 4 weeks
  Global changes in standing and active microbial communities between baseline and end of treatment as measured by beta diversity indices (Bray-Curtis and Jaccard distances).

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller CA, Corbin KD, da Costa KA, Zhang S, Zhao X, Galanko JA, Blevins T, Bennett BJ, O'Connor A, Zeisel SH. Effect of egg ingestion on trimethylamine-N-oxide production in humans: a randomized, controlled, dose-response study. Am J Clin Nutr. 2014 Sep;100(3):778-86. doi: 10.3945/ajcn.114.087692. Epub 2014 Jun 18. PMID 24944063
- [Background] Annunziata G, Maisto M, Schisano C, Ciampaglia R, Narciso V, Tenore GC, Novellino E. Effects of Grape Pomace Polyphenolic Extract (Taurisolo(R)) in Reducing TMAO Serum Levels in Humans: Preliminary Results from a Randomized, Placebo-Controlled, Cross-Over Study. Nutrients. 2019 Jan 10;11(1):139. doi: 10.3390/nu11010139. PMID 30634687
- [Background] Bergeron N, Williams PT, Lamendella R, Faghihnia N, Grube A, Li X, Wang Z, Knight R, Jansson JK, Hazen SL, Krauss RM. Diets high in resistant starch increase plasma levels of trimethylamine-N-oxide, a gut microbiome metabolite associated with CVD risk. Br J Nutr. 2016 Dec;116(12):2020-2029. doi: 10.1017/S0007114516004165. Epub 2016 Dec 20. PMID 27993177
- [Background] Cassidy A, Minihane AM. The role of metabolism (and the microbiome) in defining the clinical efficacy of dietary flavonoids. Am J Clin Nutr. 2017 Jan;105(1):10-22. doi: 10.3945/ajcn.116.136051. Epub 2016 Nov 23. PMID 27881391
- [Background] Cardona F, Andres-Lacueva C, Tulipani S, Tinahones FJ, Queipo-Ortuno MI. Benefits of polyphenols on gut microbiota and implications in human health. J Nutr Biochem. 2013 Aug;24(8):1415-22. doi: 10.1016/j.jnutbio.2013.05.001. PMID 23849454
- [Derived] Rehman A, Tyree SM, Fehlbaum S, DunnGalvin G, Panagos CG, Guy B, Patel S, Dinan TG, Duttaroy AK, Duss R, Steinert RE. A water-soluble tomato extract rich in secondary plant metabolites lowers trimethylamine-n-oxide and modulates gut microbiota: a randomized, double-blind, placebo-controlled cross-over study in overweight and obese adults. J Nutr. 2023 Jan;153(1):96-105. doi: 10.1016/j.tjnut.2022.11.009. Epub 2022 Dec 23. PMID 36913483